CLINICAL TRIAL: NCT02440490
Title: Optimising Cognitive Function in Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: The Alfred (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Katharine Baker, Katharine Baker, Monash University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CF14/2985 - 2014001639
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerised cognitive training (Experimental): The cognitive training protocol will be run using pre-validated software, HappyNeuronPro, that delivers cognitive training games. The games are designed to be visually interesting and engaging, and are varied so that each session will comprise multiple different games, to avoid boredom. They begin with easy-to-follow instructions and demonstrations, then as the participant progresses, the difficulty is automatically increased in correspondence with their performance, to avoid ceiling or plateau effects. Participants will be assigned a program targeting multiple facets of cognition found to be compromised in chronic pain states, including divided attention, working memory, mentally planning a sequence of items to form a pattern or complete a puzzle, and response inhibition.
  Interventions: Behavioral: Computerised cognitive training
- Video watching (Active Comparator): This group will be provided with a variety of videos to watch, the content of which will be in the style of documentaries on general interest topics such as nature, travel, culture, and history. Each video is followed by multiple-choice questions that participants will answer, to ensure attention was engaged. The videos are visually stimulating and engaging, but involve no increment in difficulty or requirement to improve skills. They may provide some distraction from pain and may be relaxing, interesting and informative.
  Interventions: Behavioral: Video watching

INTERVENTIONS:
Behavioral: Computerised cognitive training
  Arms: Computerised cognitive training
Behavioral: Video watching
  Arms: Video watching

SUMMARY:
Cognitive difficulties often occur with chronic pain. The aim of this randomised controlled trial is to determine whether various aspects of cognitive function can be improved. An 8-week course of cognitive training via a web-based training program (3 times per week) will be contrasted with watching informative documentary videos (for the same length of time). Outcomes include subjective and objective measures of cognition, as well as self-report measures of mood and pain.

DETAILED DESCRIPTION:
Rationale for project:

Cognitive difficulties may occur with chronic pain, potentially indicative of compromised functioning in frontal brain regions, which also results in greater difficulty controlling pain, with increased rumination and worry. Discovering a successful method for strengthening these neural systems may improve cognitive skills important for daily life and maximise therapeutic outcomes.

Research questions:

In people experiencing cognitive deficits due to their pain condition:

1. Can neurocognitive abilities be improved?
2. Can such improvements bring about better daily functioning in general?
3. If these training protocols improve cognition, will there also be an effect of pain reduction, i.e., in the extent to which pain interferes with a person's life?

Aim:

The overarching aim of this research is to determine whether cognitive function can be improved via a training protocol in people experiencing cognitive difficulties related to chronic pain.

Design:

This is a randomised controlled trial examining the effects of cognitive training compared with an active control. The investigators aim to enrol 40 participants with chronic pain in the study: 20 training, and 20 active control. This sample size was chosen based on a power analysis with moderate effect size, and is consistent with sample sizes in the existing cognitive training literature, though no similar study has so far been done in a chronic pain population. Both groups will complete their respective study activities 3 times per week, for 45 minutes each time, across 8 weeks. They will be assessed before completing the 8-week period, and again within a few days of completion.

Procedures:

40 participants will be recruited via the Caulfield Pain Management and Research Centre.

After deciding to participate and meeting all inclusion criteria, participants will be invited to attend their first on-site assessment session at Monash University, Clayton. The first assessment session will include an overview of the training program and demonstration of how to do the tasks, or an overview of the active control activities (as applicable). Both assessment sessions will involve detailed assessment of cognition, pain, and mood.

The cognitive training protocol will be run using pre-validated software that delivers brain training "games". The games are designed to be visually interesting and engaging, and are varied so that each session will comprise multiple different games, to avoid boredom. They begin with easy-to-follow instructions and demonstrations, then as the participant progresses, the difficulty is automatically increased in correspondence with their performance, to avoid ceiling or plateau effects. Participants will be assigned a program targeting multiple facets of cognition found to be compromised in chronic pain states, including divided attention, working memory, mentally planning a sequence of items to form a pattern or complete a puzzle, and response inhibition.

This software is accessible via the internet on desktop and laptop computers, or on tablet devices. All training sessions will be completed at home. The researchers will hold a master account, allowing them to log in and monitor participant progress and compliance with the training.

The active control group will be provided with a variety of videos to watch, the content of which will be in the style of documentaries on general interest topics such as nature, travel, culture, and history. These are also visually stimulating and engaging, but involve no increment in difficulty. They may provide distraction from pain and may be relaxing.

Throughout the protocol, the researchers will have weekly contact with participants by phone or video call. Keeping regular contact in this way will maintain engagement with the research team, help boost motivation and allow participants to express any issues they may be having with the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain condition
* Access to computer and internet

Exclusion Criteria:

* High dosages of opioid or benzodiazepine medication
* Currently receiving active allied health treatment
* Intellectual disability, traumatic brain injury, dementia, or other neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Objective cognitive functioning | 8 weeks
  Composite of neuropsychological test scores
Subjective cognitive functioning | 8 weeks
  Self-report measures of cognition

SECONDARY OUTCOMES:
Pain | 8 weeks
  Pain intensity and interference from the Brief Pain Inventory
Mood and coping | 8 weeks
  Self-report measures of anxiety, depression, pain catastrophizing and pain self-efficacy
Heart rate variability | 8 weeks
  Electrophysiological measure

CONTACTS AND LOCATIONS:
Overall Officials: Melita Giummarra, PhD, Principal Investigator — Monash University
Locations (1):
- Monash University, Melbourne, Australia